CLINICAL TRIAL: NCT04759183
Title: Impact of Different Virtual Reality Experiences on Anxiety and Pain
Brief Title: Virtual Reality Experiences for Anxiety and Pain Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Ryan Li, MD, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00022194; NCI-2021-00794 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00022194 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2021-02-12; First posted 2021-02-18 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Angry Birds, TRIPP) (Experimental): Patients participate in a VR intervention (Angry Birds) over 15 minutes before standard of care surgery and then participate in a VR intervention (TRIPP) over 15 minutes after surgery.
  Interventions: Other: Survey Administration; Procedure: Virtual Reality Game; Procedure: Virtual Reality Meditation
- Arm II (TRIPP, Angry Birds) (Experimental): Patients participate in a VR intervention (TRIPP) over 15 minutes before standard of care surgery and then participate in a VR intervention (Angry Birds) over 15 minutes after surgery.
  Interventions: Other: Survey Administration; Procedure: Virtual Reality Game; Procedure: Virtual Reality Meditation

INTERVENTIONS:
Other: Survey Administration — Ancillary studies
Procedure: Virtual Reality Game — Participate in VR Game "Angry Birds"
  Other Names: VR Game
Procedure: Virtual Reality Meditation — Participate in VR Meditation "TRIPP"
  Other Names: VR Meditation

SUMMARY:
This trial studies the impact of virtual reality experiences on anxiety before surgery and pain after surgery. The goal of this study is to examine how different virtual reality experiences may help reduce anxiety and improve pain control, which may help reduce the need for medications such as opioids.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To measure the impact of a gaming virtual reality (VR) experience compared to a mindfulness VR experience on preoperative anxiety and postoperative pain.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients participate in a VR intervention (Angry Birds) over 15 minutes before standard of care surgery and then participate in a VR intervention (TRIPP) over 15 minutes after surgery.

ARM II: Patients participate in a VR intervention (TRIPP) over 15 minutes before standard of care surgery and then participate in a VR intervention (Angry Birds) over 15 minutes after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older and younger than 89)
* Able to consent
* English-speaking

Exclusion Criteria:

* Non-English speaking patients because the VR content is only available in English
* Have symptoms concerning for an active respiratory infection or are on contact or isolation precautions
* Any active eye discharge
* A history of seizure, epilepsy, or hypersensitivity to flashing light
* Have a history of motion sickness or vertigo
* Have active nausea or vomiting
* Psychiatric conditions that may interfere with the ability to successfully participate in the study
* Have cardiac pacemakers
* Require hearing aids at all times that cannot be removed
* Have defibrillators
* Have wound dressings on the head or neck that prevent comfortable use of the VR headset

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
Change in preoperative anxiety scores | Baseline up to pre surgery (estimated 1 day)
  Assessed by visual analogue scale (VAS) from 0-100mm.
Change in postoperative pain scores | Baseline after surgery up to study completion (estimated 1 day)
  Assessed by VAS scale from 0-100mm.

SECONDARY OUTCOMES:
Change in blood pressure | immediately before intervention, and then immediately after intervention (estimated 1 day)
  mmHg
Patient enjoyment of each VR experience | Up to study completion (estimated 1 day)
  Likert scale (1-5). 1 represents the lowest score, and 5 represents the highest.
Change in heart rate | immediately before intervention, and then immediately after intervention (estimated 1 day)
  beats per minute (bpm)
Patient desire to use VR more in their healthcare | Up to study completion (estimated 1 day)
  Likert scale (1-5). 1 represents the lowest score, and 5 represents the highest.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan J Li, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States